CLINICAL TRIAL: NCT05483036
Title: Perception in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Alice Cronin-Golomb, Director, Vision and Cognition Laboratory, Boston University Charles River Campus
Other Study IDs: 6350X
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-08

CONDITIONS: Parkinson's Disease; Perception; Visual Hallucination
MeSH Terms: conditions — Parkinson Disease; Hallucinations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Persons with Parkinson's disease (PwPD)

SUMMARY:
The investigators plan to examine the relation of perceptual variables-basic vision, unusual perceptual experiences(including but not limited to visual hallucinations)-to relevant functional variables such as cognition, mood, and alertness/sleepiness in an online sample of persons with Parkinson's disease (PwPD). It is hypothesized that unusual perceptual experiences will relate significantly to the selected variables. Participants do not need to experience visual hallucinations to be able to participate in this study. This is an observational study only, and not an interventional study.

DETAILED DESCRIPTION:
For this study, the investigators propose to conduct an online study of PwPD (proposing a total of 60 participants) to examine the relations among variables that may relate to perception in PD. Those PwPD who express interest will be sent a link to an online survey (Qualtrics). The investigators will collect demographic and health information, followed by questionnaires assessing unusual perceptual experiences, mood, motivation, sleep, fatigue and quality of life. The survey should take roughly 45 minutes to an hour to complete.

Compensation: A $20 Amazon gift card will be offered to those who complete the survey all the way through with good effort.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 40 years old
* Have a self-reported diagnosis of idiopathic PD
* Be proficient English speakers
* Have functional vision
* Have internet access, and access to a desktop computer or laptop

Exclusion Criteria:

* Self-reported poor vision (non-functional range)
* Lack of access to internet and either a desktop computer or laptop

Ages: 40 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PwPD volunteering for an online study
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Noise Pareidolia Test | Baseline
  Assesses tendency to see meaningful objects such as faces, animals, and objects in ambiguous patterns. Higher scores (on items with no face) indicate a higher number of pareidolic responses.
Mooney Faces | Baseline
  Assesses the ability to see an upright, inverted, or scrambled face in a black and white pattern. Higher scores (on items with no face) indicate a higher number of pareidolic responses.
BU Hallucinations and Unusual Perceptual Experiences questionnaire (BU-HUPE) | Baseline
  Assesses different types of visual hallucinations - simple VH; illusions; minor hallucinations: vivid sense of presence or movement in periphery (passage); and complex VH (e.g., people, animals, objects), as well as temporal and descriptive characteristics of the hallucinations. Higher scores indicate more unusual perceptual experiences.
Prodromal Questionnaire, Brief Version (PQ-B) | Baseline
  Assesses risk for psychosis by asking about positive symptoms and related distress/impairment. Higher scores indicate higher risk for psychosis and higher related distress.
Parkinson's Disease - Psychotic Symptoms Scale (PD-PSS) | Baseline
  Assesses the frequency and severity of minor hallucinations (passage hallucinations, presence hallucinations, visual illusions), and structured hallucinations in PD. Higher scores indicate higher frequency of psychotic symptoms.
Penn Online Evaluation of Migraine (POEM) | Baseline
  Assesses headaches and migraine-related history.
Epworth Sleepiness Scale (ESS) | Baseline
  Assesses a person's general level of daytime sleepiness. Maximum Score: 24. Higher scores indicate a higher chance of dozing.
Parkinson's Disease Sleep Scale-2 | Baseline
  Assesses sleep and nocturnal disturbances in Parkinson's disease. Maximum score: 60. Higher scores indicate more frequent sleep disturbances.
Parkinson's Anxiety Scale (PAS) | Baseline
  Assesses the severity of anxiety symptoms in persons with Parkinson's disease. Maximum score:48. Higher scores indicate more severe anxiety.
Center for Epidemiological Studies Depression Scale (CES-D) | Baseline
  Assesses depressive symptoms in the general population. Maximum score:60. Higher scores indicate more severe depression.
Parkinson's Disease Questionnaire - 39 (PDQ-39) | Baseline
  Assesses Parkinson's disease-specific health-related quality of life. Higher scores indicate worse quality of life.
NIH NeuroQoL measures | Baseline
  Assesses health-related quality of life in adults with neurological disorders. Higher scores on the sub-scales indicate worse outcomes.
The Movement Disorders Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) | Baseline
  Assesses motor and non-motor experiences of daily living in Parkinson's disease. Higher scores indicate increased severity of motor and non-motor symptoms.
Non-Motor Symptoms Questionnaire (NMSQ) | Baseline
  Assesses a range of non-motor symptoms in Parkinson's disease. Higher scores indicate the presence of more non-motor symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Cronin-Golomb, PhD, Principal Investigator — Boston University
Locations (1):
- Vision and Cognition Laboratory, Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schapira AHV, Chaudhuri KR, Jenner P. Non-motor features of Parkinson disease. Nat Rev Neurosci. 2017 Jul;18(7):435-450. doi: 10.1038/nrn.2017.62. Epub 2017 Jun 8. PMID 28592904
- [Background] Barnes J, David AS. Visual hallucinations in Parkinson's disease: a review and phenomenological survey. J Neurol Neurosurg Psychiatry. 2001 Jun;70(6):727-33. doi: 10.1136/jnnp.70.6.727. PMID 11385004
- [Background] Chang A, Fox SH. Psychosis in Parkinson's Disease: Epidemiology, Pathophysiology, and Management. Drugs. 2016 Jul;76(11):1093-118. doi: 10.1007/s40265-016-0600-5. PMID 27312429
- [Background] Fenelon G, Mahieux F, Huon R, Ziegler M. Hallucinations in Parkinson's disease: prevalence, phenomenology and risk factors. Brain. 2000 Apr;123 ( Pt 4):733-45. doi: 10.1093/brain/123.4.733. PMID 10734005
- [Background] Gibson G, Mottram PG, Burn DJ, Hindle JV, Landau S, Samuel M, Hurt CS, Brown RG, M Wilson KC. Frequency, prevalence, incidence and risk factors associated with visual hallucinations in a sample of patients with Parkinson's disease: a longitudinal 4-year study. Int J Geriatr Psychiatry. 2013 Jun;28(6):626-31. doi: 10.1002/gps.3869. Epub 2012 Aug 28. PMID 22927195
- [Background] Mack J, Rabins P, Anderson K, Goldstein S, Grill S, Hirsch ES, Lehmann S, Little JT, Margolis RL, Palanci J, Pontone G, Weiss H, Williams JR, Marsh L. Prevalence of psychotic symptoms in a community-based Parkinson disease sample. Am J Geriatr Psychiatry. 2012 Feb;20(2):123-32. doi: 10.1097/JGP.0b013e31821f1b41. PMID 21617521
- [Background] Ibarretxe-Bilbao N, Ramirez-Ruiz B, Junque C, Marti MJ, Valldeoriola F, Bargallo N, Juanes S, Tolosa E. Differential progression of brain atrophy in Parkinson's disease with and without visual hallucinations. J Neurol Neurosurg Psychiatry. 2010 Jun;81(6):650-7. doi: 10.1136/jnnp.2009.179655. Epub 2009 Dec 3. PMID 19965847
- [Background] Ibarretxe-Bilbao N, Junque C, Marti MJ, Tolosa E. Cerebral basis of visual hallucinations in Parkinson's disease: structural and functional MRI studies. J Neurol Sci. 2011 Nov 15;310(1-2):79-81. doi: 10.1016/j.jns.2011.06.019. Epub 2011 Jun 25. PMID 21705027
- [Background] Goldman JG, Stebbins GT, Dinh V, Bernard B, Merkitch D, deToledo-Morrell L, Goetz CG. Visuoperceptive region atrophy independent of cognitive status in patients with Parkinson's disease with hallucinations. Brain. 2014 Mar;137(Pt 3):849-59. doi: 10.1093/brain/awt360. Epub 2014 Jan 29. PMID 24480486
- [Background] Lenka A, Jhunjhunwala KR, Saini J, Pal PK. Structural and functional neuroimaging in patients with Parkinson's disease and visual hallucinations: A critical review. Parkinsonism Relat Disord. 2015 Jul;21(7):683-91. doi: 10.1016/j.parkreldis.2015.04.005. Epub 2015 Apr 17. PMID 25920541
- [Background] Ramirez-Ruiz B, Marti MJ, Tolosa E, Gimenez M, Bargallo N, Valldeoriola F, Junque C. Cerebral atrophy in Parkinson's disease patients with visual hallucinations. Eur J Neurol. 2007 Jul;14(7):750-6. doi: 10.1111/j.1468-1331.2007.01768.x. PMID 17594330
- [Background] Goetz CG, Vaughan CL, Goldman JG, Stebbins GT. I finally see what you see: Parkinson's disease visual hallucinations captured with functional neuroimaging. Mov Disord. 2014 Jan;29(1):115-7. doi: 10.1002/mds.25554. Epub 2013 Jul 10. PMID 23843193
- [Background] Stebbins GT, Goetz CG, Carrillo MC, Bangen KJ, Turner DA, Glover GH, Gabrieli JD. Altered cortical visual processing in PD with hallucinations: an fMRI study. Neurology. 2004 Oct 26;63(8):1409-16. doi: 10.1212/01.wnl.0000141853.27081.bd. PMID 15505157
- [Background] Weil RS, Reeves S. Hallucinations in Parkinson's disease: new insights into mechanisms and treatments. Adv Clin Neurosci Rehabil. 2020 Jul 13;19(4):ONNS5189. doi: 10.47795/ONNS5189. eCollection 2020 Summer. PMID 33102741
- [Background] O'Brien J, Taylor JP, Ballard C, Barker RA, Bradley C, Burns A, Collerton D, Dave S, Dudley R, Francis P, Gibbons A, Harris K, Lawrence V, Leroi I, McKeith I, Michaelides M, Naik C, O'Callaghan C, Olsen K, Onofrj M, Pinto R, Russell G, Swann P, Thomas A, Urwyler P, Weil RS, Ffytche D. Visual hallucinations in neurological and ophthalmological disease: pathophysiology and management. J Neurol Neurosurg Psychiatry. 2020 May;91(5):512-519. doi: 10.1136/jnnp-2019-322702. Epub 2020 Mar 25. PMID 32213570
- [Background] Zhu K, van Hilten JJ, Putter H, Marinus J. Risk factors for hallucinations in Parkinson's disease: results from a large prospective cohort study. Mov Disord. 2013 Jun;28(6):755-62. doi: 10.1002/mds.25389. Epub 2013 Mar 20. PMID 23520046
- [Background] Ffytche DH, Pereira JB, Ballard C, Chaudhuri KR, Weintraub D, Aarsland D. Risk factors for early psychosis in PD: insights from the Parkinson's Progression Markers Initiative. J Neurol Neurosurg Psychiatry. 2017 Apr;88(4):325-331. doi: 10.1136/jnnp-2016-314832. PMID 28315846
- [Background] Muller AJ, Shine JM, Halliday GM, Lewis SJ. Visual hallucinations in Parkinson's disease: theoretical models. Mov Disord. 2014 Nov;29(13):1591-8. doi: 10.1002/mds.26004. Epub 2014 Aug 22. PMID 25154807
- [Background] Schwartzman D, Maravic K, Kranczioch C, Barnes J. Altered early visual processing components in hallucination-prone individuals. Neuroreport. 2008 Jun 11;19(9):933-7. doi: 10.1097/WNR.0b013e328301a640. PMID 18520996
- [Background] Archibald NK, Clarke MP, Mosimann UP, Burn DJ. The retina in Parkinson's disease. Brain. 2009 May;132(Pt 5):1128-45. doi: 10.1093/brain/awp068. Epub 2009 Mar 31. PMID 19336464
- [Background] Davidsdottir S, Cronin-Golomb A, Lee A. Visual and spatial symptoms in Parkinson's disease. Vision Res. 2005 May;45(10):1285-96. doi: 10.1016/j.visres.2004.11.006. Epub 2004 Dec 16. PMID 15733961
- [Background] Diederich NJ, Goetz CG, Raman R, Pappert EJ, Leurgans S, Piery V. Poor visual discrimination and visual hallucinations in Parkinson's disease. Clin Neuropharmacol. 1998 Sep-Oct;21(5):289-95. PMID 9789709
- [Background] Diaz-Santos M, Monge ZA, Salazar RD, Gilmore GC, Neargarder S, Cronin-Golomb A. Increasing Contrast Improves Object Perception in Parkinson's Disease with Visual Hallucinations. Mov Disord Clin Pract. 2020 Nov 17;8(1):51-59. doi: 10.1002/mdc3.13104. eCollection 2021 Jan. PMID 33426159
- [Background] Mamiya Y, Nishio Y, Watanabe H, Yokoi K, Uchiyama M, Baba T, Iizuka O, Kanno S, Kamimura N, Kazui H, Hashimoto M, Ikeda M, Takeshita C, Shimomura T, Mori E. The Pareidolia Test: A Simple Neuropsychological Test Measuring Visual Hallucination-Like Illusions. PLoS One. 2016 May 12;11(5):e0154713. doi: 10.1371/journal.pone.0154713. eCollection 2016. PMID 27171377
- [Background] Uchiyama M, Nishio Y, Yokoi K, Hosokai Y, Takeda A, Mori E. Pareidolia in Parkinson's disease without dementia: A positron emission tomography study. Parkinsonism Relat Disord. 2015 Jun;21(6):603-9. doi: 10.1016/j.parkreldis.2015.03.020. Epub 2015 Mar 31. PMID 25864093
- [Background] Murakami H, Shiraishi T, Umehara T, Omoto S, Takahashi M, Motegi H, Maku T, Sato T, Takatsu H, Komatsu T, Bono K, Sakai K, Mitsumura H, Iguchi Y. Face pareidolia is associated with right striatal dysfunction in drug-naive patients with Parkinson's disease. Neurol Sci. 2021 Dec;42(12):5327-5334. doi: 10.1007/s10072-021-05238-7. Epub 2021 Apr 22. PMID 33884529
- [Background] Watanabe H, Nishio Y, Mamiya Y, Narita W, Iizuka O, Baba T, Takeda A, Shimomura T, Mori E. Negative mood invites psychotic false perception in dementia. PLoS One. 2018 Jun 1;13(6):e0197968. doi: 10.1371/journal.pone.0197968. eCollection 2018. PMID 29856844